CLINICAL TRIAL: NCT07231237
Title: A Multi-site, Single-Arm Clinical Study Evaluating the Efficacy of Solventum™ Vitrebond™ Pulp Protect Liner/Base for Direct Capping of Pulpal Exposure Due to Trauma, Deep Caries, or Mechanical Etiology Under Dental Restorations
Brief Title: Clinical Study Evaluating Solventum™ Vitrebond™ Pulp Protect Liner/Base for Direct Capping of Pulpal Exposure
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Solventum US LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EM-11-050086
Record Dates: First submitted 2025-11-13; First posted 2025-11-17 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-11

CONDITIONS: Dental Caries; Pulp Exposure, Dental; Tooth Decay; Dental Decay
Keywords: dental; caries; cavities; pulp exposure; direct pulp capping; Vitrebond Pulp Protect; pulp vitality; dentin bridge; pulp protection
MeSH Terms: conditions — Dental Caries; Dental Pulp Exposure

STUDY DESIGN:
Intervention Model Description: Multi-site, single arm clinical study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Vitrebond™ Pulp Protect Liner/Base (Experimental): Vitrebond™ Pulp Protect Liner/Base used for Direct Pulp Capping
  Interventions: Device: Vitrebond™ Pulp Protect Liner/Base

INTERVENTIONS:
Device: Vitrebond™ Pulp Protect Liner/Base — Vitrebond™ Pulp Protect Liner/Base used for Direct Pulp Capping

SUMMARY:
This research study is looking at the safety and effectiveness of Solventum™ Vitrebond™ Pulp Protect Liner/Base for direct pulp capping (DPC) on permanent teeth that have pulp exposure due either to deep cavities, trauma, or other accidental causes. Dental pulp is the part of the tooth that contains the nerves, blood vessels, and cells that keep teeth healthy. The DPC procedure is done by dentists to help preserve tooth health if there is pulp exposure during the tooth restoration or due to trauma. Participants must have at least one permanent tooth with pulp exposure that needs DPC to be eligible for the study.

DETAILED DESCRIPTION:
This is a multi-site, single-arm, prospective clinical study evaluating Solventum™ Vitrebond™ Pulp Protect Liner/Base treatment for direct pulp capping on permanent teeth. Vitrebond™ Pulp Protect Liner/Base is a new product designed to be placed under dental fillings that can be used as a "Liner/Base" to create a lining between the tooth and the filling to reduce sensitivity, and for direct pulp capping if there is a small amount of dental pulp exposed during the restoration.

The purpose of this clinical study will be to assess the effectiveness and safety of Vitrebond™ Pulp Protect for direct pulp capping on permanent teeth that have pulp exposure due either to deep cavities, trauma, or other accidental causes. The primary objective is to evaluate Vitrebond™ Pulp Protect Liner/Base in maintaining pulp vitality (a measure of tooth health) when used for pulp capping, measured at 1-year post-restoration. The secondary objective of this study is to evaluate treated teeth for abnormal clinical signs or symptoms for up to 5 years after treatment to assess long-term safety and effectiveness. The success of Vitrebond™ Pulp Protect for direct pulp capping in this single-arm clinical study will be determined based on an assessment of pulp vitality one year after restoration compared to a pre-specified performance goal derived from literature using calcium hydroxide as the reference comparator.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is age 7 years or older at time of consent.
2. Subject is in good general health (i.e., meets American Society of Anesthesiologists (ASA) Level I or ASA Level II classification criteria).
3. Subject or Subject's Legally Authorized Representative is able and willing to understand and sign an Informed Consent Form or give Assent, as applicable.
4. Subject is able and willing to return in-person for all scheduled study visits.
5. Subject is able and willing to follow study restrictions.
6. Subject has existing dental radiographic images of the study teeth of current and acceptable diagnostic quality taken within 3 months of tooth restoration.
7. Study tooth has healthy periodontal tissues or mildly inflamed tissues not associated with trauma, with probing depths no greater than 4 mm and no gingival recession associated with self-reported sensitivity.
8. Study tooth has no pre-operative sensitivity or exhibit pre-operative sensitivity that is relieved immediately after stimulus removal.
9. Study tooth has a positive response to a sensibility test (i.e., cold test using a refrigerant spray).
10. Study tooth can be restored with a direct permanent restoration (stepwise caries removal will not be used).
11. Study teeth are on opposite right/left sides of the mouth (for Subjects with more than one candidate study tooth).
12. Study tooth will be restored no later than 1 month after the date of the first study tooth's restoration (for Subjects with more than one candidate study tooth).

    Intra-operative Inclusion Criteria:
13. Subject has one or more permanent teeth with pinpoint pulpal exposure (0.5 mm - 1.0 mm in diameter) needing direct pulp capping, excluding third molars.

Exclusion Criteria:

1. Subject has a history of adverse reaction to any materials used in this study, including but not limited to acrylates.
2. Subject is unable, for any reason, to tolerate the study procedures (e.g., use of a rubber dam) or the length of time required to complete the restoration(s) on the study tooth/teeth.
3. Subject is taking part in or planning to be enrolled in a clinical evaluation of any other dental materials at any time during the study.
4. Subject has a history of chronic use of anti-inflammatory, analgesic (pain), and/or mind-altering drugs for medical (including psychiatric) and pharmacotherapeutic therapies that might alter perception of pain.
5. Subject is pregnant or breast feeding at the time of screening.
6. Subject has any spontaneous or other orofacial pain (excluding pain from trauma cases, which may exhibit spontaneous pain due to tooth fracture) within the same quadrant as the study tooth that may interfere with assessment of sensitivity.
7. Study tooth diagnosed with cracked tooth syndrome.
8. Study tooth mobility >= grade 2 using the Miller's tooth mobility index.
9. Study tooth has previous and current signs and symptoms of pulpal and/or periapical disease (e.g., root resorption or pulpal calcifications) or irreversible pulpitis (excluding pain from trauma cases).
10. Study tooth has no systemic mineralization pathology (e.g., amelogenesis imperfecta, enamel hypoplasia, etc.)
11. Study tooth that is not restorable
12. Study tooth that requires a crown preparation.
13. Subject is, in the opinion of the Investigator, unsuitable for enrollment in the study for reasons other than those specified in the above exclusion criteria.
14. Study tooth has an existing restoration or requires a new restoration that interferes with radiographic assessments (e.g., caries on the buccal surface).

    Intra-operative Exclusion Criteria:
15. Study tooth exhibits bleeding of the exposed pulp that does not stop within 8 minutes.

Ages: 7 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 350 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2027-12 (Estimated); Study Completion 2032-02 (Estimated)

PRIMARY OUTCOMES:
Pulp Vitality at 1-year | 1 year post-restoration
  Pulp vitality, assessed by pulp sensibility testing using a refrigerant spray intended for dental use. A positive response from the pulp sensibility test is indicative of the pulp vitality of the tooth (primary endpoint).
  Categories for pulp vitality will include:
  1. Vital pulp (normal): Positive response from the pulp sensibility test that subsides within 5 seconds.
  2. Reversible pulpitis: Positive response from pulp sensibility test that lasts greater than 5 seconds up to approximately 30 seconds.
  3. Irreversible pulpitis: Prolonged positive response from pulp sensibility test that lasts more than approximately 30 seconds.
  4. Non-vital pulp: Negative response from the pulp sensibility test.

SECONDARY OUTCOMES:
Pulp Vitality at baseline, 3 months, 6 months, and 2, 3, 4, and 5 years | Baseline, 3 months, 6 months, and 2, 3, 4, and 5 years post-restoration.
  Pulp vitality, assessed by pulp sensibility testing using a refrigerant spray intended for dental use. A positive response from the pulp sensibility test is indicative of the pulp vitality of the tooth (primary endpoint).
  Categories for pulp vitality will include:
  1. Vital pulp (normal): Positive response from the pulp sensibility test that subsides within 5 seconds.
  2. Reversible pulpitis: Positive response from pulp sensibility test that lasts greater than 5 seconds up to approximately 30 seconds.
  3. Irreversible pulpitis: Prolonged positive response from pulp sensibility test that lasts more than approximately 30 seconds.
  4. Non-vital pulp: Negative response from the pulp sensibility test.
Reparative dentin formation | 6 months and 1 year, and only if taken at the 2-, 3-, 4-, and 5-year post-restoration
  Signs of reparative dentin formation assessed by bitewing (for posterior teeth) or periapical (for anterior teeth) radiographs taken at scheduled follow-up visits. Reparative dentin formation is desired.
  Categories for reparative dentin formation will include:
  1. Presence of reparative dentin formation
  2. Absence of reparative dentin formation
Apical periodontitis | 6-months and 1-year post-restoration, and at 2-, 3-, 4-, and 5-years post-restoration if periapical radiographs are taken
  Apical periodontitis will be assessed by the clinician based on clinical assessments of symptoms (percussion of teeth, palpation of nearby bone, and visual examination of tissues) as well as periapical radiographs taken at scheduled follow-up visits. Absence of apical periodontitis is desired.
  Categories for apical periodontitis (symptomatic and/or asymptomatic) formation will include:
  1. Presence of apical periodontitis
  2. Absence of apical periodontitis
Internal root resorption | 6 months and 1 year, and if taken at the 2-, 3-, 4-, and 5-years post-restoration
  Internal root resorption will be assessed by periapical radiographs taken at each scheduled follow-up visit at 6 months and 1 year, and if taken at the 2-, 3-, 4-, and 5-year follow-up visits and any unscheduled visits involving study teeth. Absence of internal root resorption is desired.
  Categories for internal root resorption will include:
  1. Presence of internal root resorption
  2. Absence of internal root resorption
External root resorption | 6 months and 1 year, and if taken at the 2-, 3-, 4-, and 5-years post-restoration
  External root resorption will be assessed by periapical radiographs taken at each scheduled follow-up visit at 6 months and 1 year, and if taken at the 2-, 3-, 4-, and 5-year follow-up visits and any unscheduled visits involving study teeth. Absence of external root resorption is desired.
  Categories for external root resorption will include:
  1. Presence of external root resorptions
  2. Absence of external root resorptions
Pulp canal obliteration | 6 months and 1 year, and if taken at the 2-, 3-, 4-, and 5-years post-restoration
  Pulp canal obliteration will be assessed by periapical radiographs taken at each scheduled follow-up visit at 6 months and 1 year, and if taken at the 2-, 3-, 4-, and 5-year follow-up visits and any unscheduled visits involving study teeth. Absence of pulp canal obliteration is desired.
  Categories for pulp canal obliteration will include:
  1. Presence of pulp canal obliteration
  2. Absence of pulp canal obliteration
Pathological tooth mobility | baseline, 3 months, 6 months, and 1, 2, 3, 4, and 5 years post-restoration
  Pathological tooth mobility will be assessed by clinicians at scheduled visits. The American Academy of Periodontology definition of tooth mobility is the movement of a tooth in its socket resulting from an applied force.
  Categories for pathological tooth mobility using the Miller's tooth mobility index will include:
  1. Class 0: normal (physiologic) movement when force is applied
  2. Class 1: < 1 mm (horizontal)
     a. mobility greater than physiologic
  3. Class 2: ≥1 mm (horizontal),
     1. tooth can be moved 1 mm or more in a lateral direction (buccolingual or mesiodistal); and
     2. inability to depress the tooth in a vertical direction (apicocoronal)
  4. Class 3: ≥1 mm (horizontal and vertical)
     1. tooth can be moved 1 mm or more in a lateral direction (buccolingual or mesiodistal); and
     2. ability to depress the tooth in a vertical direction (apicocoronal)
Spontaneous pain | baseline, 3 months, 6 months, and 1, 2, 3, 4, and 5 years post-restoration
  Spontaneous pain not due to a stimulus will be self-assessed by subjects for each study tooth at scheduled visits. The baseline spontaneous pain assessment should be conducted a minimum of 3 hours after completing the restoration to allow time for the anesthesia to wear off. The baseline assessment may be conducted via phone to ask the subject if they are experiencing any spontaneous pain in the study tooth and must be completed within 1 week of the tooth restoration. The absence of spontaneous pain is desired.
  Spontaneous pain is defined as prolonged intense pain that doesn't respond to over-the-counter pain medication, and/or pain that wakes you up from sleep.
  Categories for spontaneous pain will include:
  1. Presence of spontaneous pain
  2. Absence of spontaneous pain

CONTACTS AND LOCATIONS:
Overall Officials: Mabi Singh, DMD, BDS, MS, Principal Investigator — Tufts University
Locations (1):
- Tufts University, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Miller, S.C, Textbook of periodontia, Blakiston Company, Philidelphia, 1938